CLINICAL TRIAL: NCT03678792
Title: Time to Detox: A Patient-Centered Comparison of Length of Detoxification Treatment and Time to Naltrexone Maintenance Therapy in Opioid-Dependent Individuals
Brief Title: Comparison of Three Opioid Detoxification Treatment Regimens
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Infeasible to conduct at this time.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Cropsey, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001612
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Opioid-Related Disorders; Opioid Withdrawal
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Morphine; Tramadol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Buprenorphine-Naloxone (Other): Standard of Care
  Interventions: Drug: Buprenorphine/naloxone
- Morphine (Experimental)
  Interventions: Drug: Morphine
- Tramadol (Experimental)
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Participants in this group will be tapered on buprenorphine-naloxone regimen, 2mg/day
  Arms: Buprenorphine-Naloxone
Drug: Morphine — Participants in this group will be tapered on an oral morphine regimen, 30-60mg/day
  Arms: Morphine
Drug: Tramadol — Participants in this group will be tapered on an oral morphine regimen, 50-100mg/day
  Arms: Tramadol

SUMMARY:
Despite an increased focus on treating opioid use disorder there are relatively few studies that compare the length of time required for detoxification with medications other than buprenorphine. Morphine and tramadol have shorter half-lives than buprenorphine and can be used for opioid detoxification. The proposed protocol aims to address this gap by directly comparing the length of treatment required for detoxification from opioids in a patient-centered manner with oral morphine, tramadol, or buprenorphine-naloxone as well as comparing the severity of withdrawal experienced by patients in each group. The investigators predict that treatment with oral morphine or tramadol will result in a faster completion of detoxification and initiation of naltrexone maintenance.

DETAILED DESCRIPTION:
Opioid dependent individuals will be recruited for participation in the study. Upon recruitment into the randomized trial each participant will be started on an induction dosage of medication intended to suppress withdrawal (either buprenorphine-naloxone, morphine, or tramadol). Participants will remain on the induction dose for at least 24 hrs. Severity of withdrawal will be assessed twice a day using the Clinical Opiate Withdrawal Scale (COWS) and the Subjective Opiate Withdrawal Scale (SOWS). Each morning, participants will be given the option to progress on the tapering protocol (see below for individual regimens). Time to complete detoxification and initiation of naltrexone treatment will be measured. At completion of the study each participant will complete a 7-iten Detoxification Treatment Satisfaction questionnaire.

Taper Schedule Dosing Buprenorphine-Naloxone (Suboxone): Patients will get 4mg when withdrawal symptoms start. Patients can receive the first 8mg dose as early as 6hrs later, and at that point will start on an 8mg twice-a-day schedule. Each morning the patient will be assessed regarding their ability to progress to the next stage of the taper. Buprenorphine-naloxone will be tapered 2mg/day.

Tramadol: At enrollment the patients will receive a 100mg dose and can receive another 100mg every 6 hrs for 24 hrs. Each morning the patient will be assessed regarding their ability to progress to the next stage of the taper. Patients will then be tapered on the following schedule 100mg every 8 hrs, 50mg every 6 hrs, 50mg every 8 hrs, 50mg ever 12 hrs, and one final daily dose of 50mg.

Morphine: Patients receive 30mg every 4 hours for 24 hrs from when withdrawal symptoms start. Each morning the patient will be assessed regarding their ability to progress to the next stage of the taper. Patients will then be tapered on the following schedule: 30 mg every 6 hours, 30 mg every 8 hours, 30 mg every 12 hours, and one final daily 30 mg dose.

As Needed Medications: Patients in all groups will have access to the following medications as needed gabapentin 400mg every 8 hrs, loperamide 2mg every 3 hrs, odansetron 4mg every 6 hrs, ibuprofen 600mg ever 8 hrs, and hydroxyzine 25-50mg nightly.

Naltrexone Test Dose Patients will receive an oral test dose of naltrexone (25mg) either 10 days after completing the buprenorphine-naloxone taper (standard of care) or 7 days after the morphine or tramadol taper. If the oral test dose is tolerated then the patients may choose to pursue treatment with an extended release naltrexone intramuscular injection (380mg) 24 hrs later. Due to the risk for hepatocellular injury with naltrexone, patients with baseline elevations in either aspartate transaminase or alanine transaminase greater than three times the upper limit of our clinical laboratory's reference range will be ineligible to receive extended release naltrexone, but may choose to continue oral naltrexone maintenance therapy (50mg daily) (standard of care). As part of the study the investigators will record the time to naltrexone maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Meeting DSM-V criteria for opioid use disorder
* Current use of opiates
* Displaying evidence of opioid withdrawal
* Having no significant current medical/psychiatric illness
* English speaking

Exclusion Criteria:

* Use of methadone or buprenorphine exclusively
* Pregnancy
* Hypotensive
* History of seizures
* Physical dependence on alcohol and/or benzodiazepines that requires treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-15 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10-25 (Estimated)

PRIMARY OUTCOMES:
Time to detoxification regimen completion | Five to twenty days
  Will be measured from first to last dose of tapering medication
Time to naltrexone test dose | 12 to 30 days
  Measured from first dose of tapering medication to naltrexone test dose

SECONDARY OUTCOMES:
Subjective Opiate Withdrawal Scale | Five to twenty days
  The Subjective Opiate Withdrawal Scale (SOWS) measures the severity of 16 symptoms of opiate withdrawal as rated by the patient on a scale of 0 (not at all) to 4 (extremely). Total scores for each patient will be recorded each day and compared between treatment groups.
Clinical Opiate Withdrawal Scale | Five to twenty days
  The Clinical Opiate Withdrawal Scale (COWS) measures the severity of 11 signs and symptoms of opiate withdrawal as rated by a healthcare provider. Each symptom is rated 0 (either no symptom or abnormal sign present) to 4 or 5 (sign or symptom is prominent or severe). Scores are considered severe if greater than 36, moderately severe if 25-36, moderate if 13-25, and mild if 5-12. Maximum score possible is 48. Total scores across treatment will be compared between treatment groups.
Total use of 'as needed medications' during detoxification | Five to twenty days
  The following medications will be available to all patients throughout the the study; gabapentin, loperamide, ondansetron, ibuprofen, and hydroxyzine. The total amount of these 'as needed' medications will be recorded and compared between the different treatment groups.
Treatment Satisfaction Survey | One day
  To assess treatment satisfaction each patient will complete a 6-question survey at the end of the study protocol. Patients will be asked to rate their satisfaction with their medication treatment, from very dissatisfied to very satisfied, how bothersome withdrawal symptoms were, from very bothersome to not at all bothersome, what if any side effects were experience, and by how much the medication reduced cravings, from not at all to completely.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Florence CS, Zhou C, Luo F, Xu L. The Economic Burden of Prescription Opioid Overdose, Abuse, and Dependence in the United States, 2013. Med Care. 2016 Oct;54(10):901-6. doi: 10.1097/MLR.0000000000000625. PMID 27623005
- [Background] Jiang R, Lee I, Lee TA, Pickard AS. The societal cost of heroin use disorder in the United States. PLoS One. 2017 May 30;12(5):e0177323. doi: 10.1371/journal.pone.0177323. eCollection 2017. PMID 28557994
- [Background] Mattick RP, Breen C, Kimber J, Davoli M. Buprenorphine maintenance versus placebo or methadone maintenance for opioid dependence. Cochrane Database Syst Rev. 2014 Feb 6;2014(2):CD002207. doi: 10.1002/14651858.CD002207.pub4. PMID 24500948
- [Background] Skeie I, Brekke M, Gossop M, Lindbaek M, Reinertsen E, Thoresen M, Waal H. Changes in somatic disease incidents during opioid maintenance treatment: results from a Norwegian cohort study. BMJ Open. 2011 Aug 6;1(1):e000130. doi: 10.1136/bmjopen-2011-000130. PMID 22021771
- [Background] Bukten A, Roislien J, Skurtveit S, Waal H, Gossop M, Clausen T. A day-by-day investigation of changes in criminal convictions before and after entering and leaving opioid maintenance treatment: a national cohort study. BMC Psychiatry. 2013 Oct 16;13:262. doi: 10.1186/1471-244X-13-262. PMID 24131480
- [Background] Comer SD, Sullivan MA, Yu E, Rothenberg JL, Kleber HD, Kampman K, Dackis C, O'Brien CP. Injectable, sustained-release naltrexone for the treatment of opioid dependence: a randomized, placebo-controlled trial. Arch Gen Psychiatry. 2006 Feb;63(2):210-8. doi: 10.1001/archpsyc.63.2.210. PMID 16461865
- [Background] Sullivan M, Bisaga A, Pavlicova M, Choi CJ, Mishlen K, Carpenter KM, Levin FR, Dakwar E, Mariani JJ, Nunes EV. Long-Acting Injectable Naltrexone Induction: A Randomized Trial of Outpatient Opioid Detoxification With Naltrexone Versus Buprenorphine. Am J Psychiatry. 2017 May 1;174(5):459-467. doi: 10.1176/appi.ajp.2016.16050548. Epub 2017 Jan 10. PMID 28068780
- [Background] Fishbain DA, Rosomoff HL, Cutler R. Opiate detoxification protocols. A clinical manual. Ann Clin Psychiatry. 1993 Mar;5(1):53-65. doi: 10.3109/10401239309148924. PMID 8394176
- [Background] Threlkeld M, Parran TV, Adelman CA, Grey SF, Yu J. Tramadol versus buprenorphine for the management of acute heroin withdrawal: a retrospective matched cohort controlled study. Am J Addict. 2006 Mar-Apr;15(2):186-91. doi: 10.1080/10550490500528712. PMID 16595358
- [Background] Zarghami M, Masoum B, Shiran MR. Tramadol versus methadone for treatment of opiate withdrawal: a double-blind, randomized, clinical trial. J Addict Dis. 2012;31(2):112-7. doi: 10.1080/10550887.2012.665728. PMID 22540433
- [Background] Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003 Apr-Jun;35(2):253-9. doi: 10.1080/02791072.2003.10400007. PMID 12924748
- [Background] Handelsman L, Cochrane KJ, Aronson MJ, Ness R, Rubinstein KJ, Kanof PD. Two new rating scales for opiate withdrawal. Am J Drug Alcohol Abuse. 1987;13(3):293-308. doi: 10.3109/00952998709001515. PMID 3687892
- See also: Behavioral health trends in the United States: Results from the 2014 National Survey on Drug Use and Health — https://www.samhsa.gov/data/sites/default/files/NSDUH-FRR1-2014/NSDUH-FRR1-2014.pdf